CLINICAL TRIAL: NCT02201849
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Oral ALKS 8700 in Healthy Adults
Brief Title: A Study of ALKS 8700, a Monomethyl Fumarate (MMF) Molecule, in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK8700-001
Record Dates: First submitted 2014-07-18; First posted 2014-07-28 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis
Keywords: Alkermes; ALKS 8700
MeSH Terms: conditions — Multiple Sclerosis | interventions — Drug Evaluation; Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study Drug (Experimental): Oral capsules
  Interventions: Drug: Study Drug
- Active Control (Active Comparator): Oral capsules
  Interventions: Drug: Active Control
- Placebo (Placebo Comparator): Oral capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Study Drug
  Other Names: ALKS 8700 capsules
  Arms: Study Drug
Drug: Active Control
  Other Names: TECFIDERA® capsules
  Arms: Active Control
Drug: Placebo
  Other Names: Placebo capsules
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of ALKS 8700, a monomethyl fumerate (MMF) molecule.

DETAILED DESCRIPTION:
This study record was previously posted/updated by Alkermes, Inc. As of 29 Oct 2019, the sponsorship of the trial was transferred to Biogen along with responsibility for subsequent updates to the record.

ELIGIBILITY:
Inclusion Criteria:

* Has a body-mass Index (BMI) >/=18.0 and </=32.0 kg/m2
* Agrees to use an acceptable method of contraception for the duration of the study and for 30 days after any study drug administration
* Additional criteria may apply

Exclusion Criteria:

* Is currently pregnant or breastfeeding
* Has a lifetime history of menopausal hot flashes
* Has a clinically significant medical condition
* Has had a clinically significant illness in the 30 days prior to first study drug administration
* Has had a serious infection (eg, pneumonia or septicemia) within the 3 months prior to study drug administration
* Has had any vaccinations in the 4 weeks prior to inpatient admission
* Has a lifetime history of diabetes
* Additional criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be measured by incidence of adverse events | up to 27 days

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | up to 27 days
  Concentrations will be measured predose and at 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3, 4, 6, 8, 10, 12, 24, 36, 48, and 72 hours postdose
Time to attain Cmax (Tmax) | Up to 27 days
Area under the concentration-time curve from 0 to the last quantifiable time interval (AUClast) | Up to 27 days
Area under the concentration-time curve from time 0 to infinity (AUCinf) | Up to 27 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Alkermes Investigational Site, Austin, Texas, United States